CLINICAL TRIAL: NCT01943812
Title: Substituted Frozen Embryo Transfer Cycles With GnRH-agonist Supplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Humaidan (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, D.M.Sc., M.D., Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skive-2013-BA
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Pregnancy Loss; Frozen Embryo Transfer
MeSH Terms: interventions — Estradiol; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Substituted FET cycle and GnRHa (Experimental): Substituted FET GnRH-a 2 bolus two days before Estradiol 6 mg Progesterone (Crinone) 180 mg
  Interventions: Drug: Estradiol and progeterone
- Substituted FET cycle (Active Comparator): substituted FET cycle Estradiol Progesterone
  Interventions: Drug: Estradiol and progeterone

INTERVENTIONS:
Drug: Estradiol and progeterone — Estradiol and progesterone
  Other Names: Estradiol and progesterone

SUMMARY:
The aim of this study is to compare two FET protocols by modifying the substituted FET cycle in order to maintain a higher ongoing positive pregnancy rate and thus reduce the early pregnancy loss.

Hypothesis: adding GnRH-agonist to the substituted cycle in FET treatment reduces the early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial thickness ≥ 7 mm after stimulation
* 18-45 years
* IVF/ICSI fertilisation
* BMI > 18,5 <30 kg/m2
* cycle length 25-34 days

Exclusion Criteria:

* endometrial thickness < 7 mm or no triple layer endometrium and/or functional follicles
* Uterine abnormality
* Chronic medical disease
* oocyte donation cycles

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 287 (Actual)
Dates: Start 2013-12; Primary Completion 2019-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Pregnancy loss rate | Primary outcome is avaible after 12th week of gestational.

SECONDARY OUTCOMES:
Pregnancy rate | 14 days after embryo transfer.

OTHER OUTCOMES:
Luteal progesterone levels | 7th week of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Alsbjerg, M.D., Principal Investigator — Fertility Clinic Regional Hospital Skive
Locations (2):
- Denmark (2):
  - IVF syd, Fredericia
  - Fertility Clinic Regional Hospital Skive, Skive